CLINICAL TRIAL: NCT02812212
Title: Cortical Transit Time on Diuretic Renogram as an Early Marker of Significant Obstruction in Antenatally Detected Uretero-pelvic Junction Syndrome
Brief Title: CTT on Renogram as an Early Marker of Significant Obstruction in Uretero-pelvic Junction Syndrome
Acronym: JUMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/CHU/11
Record Dates: First submitted 2016-06-17; First posted 2016-06-24 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Ureteropelvic Junction Obstruction
Keywords: ureteropelvic junction obstruction; cortical transit time
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label (Experimental): Device: ultrasonography and diuretic renography Bilateral ultrasonography to measure the antero-posterior renal pelvic diameter (APRPD) in both positions.
  Diuretic renography to measure the cortical transit time
  Interventions: Device: ultrasonography; Device: diuretic renography

INTERVENTIONS:
Device: ultrasonography — bilateral ultrasonography to measure the antero-posterior renal pelvic diameter (APRPD) in both positions.
Device: diuretic renography — diuretic renography to measure the cortical transit time.

SUMMARY:
Cortical transit time on diuretic renogram as an early marker of significant obstruction in antenatally detected uretero-pelvic junction syndrome

DETAILED DESCRIPTION:
Antenatal hydronephrosis (ANH) is an uropathy characterized by a dilatation of the renal collecting system. It is the most common abnormality found during prenatal ultrasound examination (1-5% pregnancies). Though the majority of cases are transient or "functional" and ultimately resolve after birth, some cases have a pathological origin of which ureteropelvic junction obstruction (UPJO) is the most common (7-35% cases).

An increased understanding of the natural history of ANH has been accompanied by a change in its management from systematic surgical approach to active surveillance and selective surgery. The main challenge is then to differentiate reversible ANH from pathological UPJO. Pathological obstruction generally results in an impairment of urine flow which, if left untreated, will result in renal damage or abnormal development of the kidney. It is therefore up to the paediatric urologist to determine whether the obstruction is significant before any irreversible damage occurs. However, without reliable prognostic criteria identified to date, controversy still exists regarding the indication and optimal timing for surgical management of UPJO.

Diuretic renography is currently the most widely used diagnostic modality to evaluate renal function and obstruction. It confirms significant obstruction when it demonstrates alteration of renal function, but having to wait for significant and potentially irreversible loss of function to be able to confirm surgical indication is unsatisfactory.

For many authors increase in hydronephrosis, defined as an increase in the dilatation of antero-posterior renal pelvic diameter (APRPD), is a marker of significant obstruction. But again, having to wait for an increase in hydronephrosis, which is by definition deterioration of the kidney, even if it precedes loss of function, remains unsatisfactory and therefore an earlier marker is needed to improve patients' management.

Determining a reliable early predictive marker for future deterioration of renal function in children with UPJO will considerably change current management of these children by avoiding unnecessary surgery for reversible cases and by being able to offer early surgery before renal deterioration for pathological cases. It could also determine which patients need close surveillance and which do not need to be monitored as often.

Two potential markers have been recently described: the cortical transit time (CTT) measured on renogram, which was shown in a recent retrospective study, to be associated with the need or not for surgery, and positional variation in APRPD as measured by sonography, which was also found to have prognostic value in a recently published pilot study. Both criteria are promising but need to be evaluated prospectively in larger population.

The investigators propose to study prospectively the prognostic value of CTT and as a secondary objective, to determine the prognostic value of positional variation in APRPD. The investigators will then be able to compare these two prognostic markers.

ELIGIBILITY:
Inclusion Criteria:

Infants:

* Aged of 4 to 8 weeks of life
* Presenting an ureteropelvic junction obstruction (UPJO) detected before birth by ultrasound
* Presenting an UPJO, defined by an Antero-Posterior Renal Pelvic Diameter greater or equal to 15 mm, confirmed by ultrasound post-natally between the 1st and 15th day of life
* Presenting a unilateral UPJO
* whose legal representatives have provided a signed free and informed written consent for their infant's participation
* whose at least one of his legal representative is affiliated to national social security

Exclusion Criteria:

Infants presenting:

* A bilateral UPJO
* An ureteral dilatation
* An associated contralateral uropathy
* A solitary kidney
* A renal insufficiency
* Severe associated disabilities ( ie polymalformation syndromes)
* A concomitant participation in another trial
* A contraindication to furosemide (acute renal insufficiency, hepatic encephalopathy, hypovolemia or dehydration, severe hypokalemia, severe hyponatremia)
* A contraindication to the radionuclide marker (hypersensitivity to the active substance or to excipients)

Ages: 4 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
risk, during the first year of life, of an increase of 4mm or more in the measure of APRPD by ultrasonography as compared to the baseline measure, according to the presence or not of an abnormal cortical transit ti | 3 months, 6 months and 12 months
  During the first year of life, the antero-posterior renal pelvic diameter will be measured by ultrasonography at baseline, then at 3 months, 6 months and 12 months after baseline.
  Diuretic renography will be performed only at baseline and the cortical transit time will be classified as normal or abnormal.
  An increase of 4mm or more of APRPD is the threshold chosen in the study to determine the aggravation of hydronephrosis.
  The occurence of the increase of 4mm or more in the measure of APRPD will be compared with the normality/abnormality of the cortical transit time in order to determine its value as a prognostic marker.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Harper, MD, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - CHU de Bordeaux, Bordeaux
  - CHU de Limoges, Limoges
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes
  - Centre Hospitalier Universitaire de La Réunion, Saint-Denis

IPD SHARING:
Plan to Share IPD: No